CLINICAL TRIAL: NCT02744651
Title: EUS-Endodrill vs. EUS-FNA for Diagnosis of Submucosal Tumors in the Upper GI Tract
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Practical circumstances making it not possible to finish the study.
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Martin Jeremiasen, Consultant Surgeon, Region Skane
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Endodrill III
Record Dates: First submitted 2016-04-05; First posted 2016-04-20 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Gastrointestinal Neoplasms
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-FNA (Active Comparator): All patients with a confirmed suspicion of a submucosal tumor in the upper GI tract will be included in this study. A senior endoscopist will perform multiple passes of EUS-FNA until she/he has collected enough material for the pathologist to establish a possible diagnosis.
  Interventions: Device: EUS-FNA
- EUS-Endodrill biopsy (Active Comparator): All patients who are included in the study will also be examined by a senior endoscopist performing multiple EUS guided passes with the Endodrill biopsy. The harvested tissue from the tumor will be examined by a pathologist in order to establish a diagnosis.
  Interventions: Device: EUS-Endodrill biopsy

INTERVENTIONS:
Device: EUS-FNA — Please note the text in section "Arm description"
  Arms: EUS-FNA
Device: EUS-Endodrill biopsy — Please note the text in section "Arm description"
  Arms: EUS-Endodrill biopsy

SUMMARY:
Endodrill is a new instrument for biopsy sampling in the GI-channel. The purpose of this study is as follows:

- Compare EUS-guided Endodrill biopsies with endoscopic ultrasound guided fine needle aspiration (EUS-FNA) in terms of ability to establish the correct diagnosis of submucosal tumors in the upper GI tract.

DETAILED DESCRIPTION:
Endodrill is a newly constructed biopsy tool for flexible endoscopic use. It uses a drilling motion within a casing to harvest solid biopsies from tissue through the biopsy channel of a conventional flexible endoscope. It was originally designed for sampling of tissue from submucosal lesions. The investigators first study of the instrument is now finished. Endodrill is safe to use and generates more submucosal tissue compared to biopsies with a conventional biopsy forceps.

In this study the investigators want to compare the Endodrill instrument with FNA (both modalities EUS-guided) in terms of ability to obtain the correct diagnosis of submucosal tumors in the upper GI-tract. Patients diagnosed with suspected submucosal tumors in the upper GI-tract will be enrolled to this study. They will first go through examination with EUS. If the suspicion of a submucosal tumor is confirmed, the investigator will perform both EUS guided FNA and Endodrill biopsies in the same patient.The harvested tissue will be evaluated by senior pathologists to clarify which method that generates most correct diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a suspected submucosal tumor in the upper GI tract that are available for both EUS-guided FNA and Endodrill biopsy

Exclusion Criteria:

* Mental illness
* Extreme co-morbidity

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of correct histopathological diagnoses from submucosal tumors in the upper GI tract. | 24 months
  Number of biopsies with the correct histopathological diagnoses

CONTACTS AND LOCATIONS:
Overall Officials: Jan Johansson, SrConsultant, Principal Investigator — Region Skåne
Locations (1):
- University Hospital of Lund, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No